CLINICAL TRIAL: NCT03255824
Title: A Comparison of Dexmedetomidine Versus Propofol for Use in Intravenous Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Nolan, Attending Oral Maxillofacial Surgery, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2016-6953
Record Dates: First submitted 2017-06-28; First posted 2017-08-21 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Anesthesia
Keywords: Oral Surgery; Third Molars; Intravenous Sedation; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Propofol; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propofol Group (Active Comparator): Group of patients to be administered a standard Propofol, Midazolam, Fentanyl anesthesia combination.
  Interventions: Drug: Propofol, Midazolam, and Fentanyl
- Dexmedetomidine Group (Experimental): Group of patients to be administered the Dexmedetomidine and Midazolam anesthesia combination.
  Interventions: Drug: Dexmedetomidine and Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine and Midazolam — Administration of Dexmedetomidine and Midazolam for sedation during third molar surgery.
  Other Names: Precedex
  Arms: Dexmedetomidine Group
Drug: Propofol, Midazolam, and Fentanyl — Administration of Propofol, Midazolam, and Fentanyl for sedation during third molar surgery.
  Other Names: Diprivan
  Arms: Propofol Group

SUMMARY:
Hypothesis: A combination of midazolam with dexmedetomidine for sedation during third molar surgery will provide 1) superior patient satisfaction, 2) superior operator satisfaction and 3) no significant hemodynamic or respiratory changes when compared to a sedation combination of midazolam, fentanyl and propofol for sedation during third molar surgery.

DETAILED DESCRIPTION:
Intravenous sedation (IVS) is an integral aspect of the oral and maxillofacial surgeon's practice. For many minor oral surgical procedures, intravenous sedation is often necessary to manage patient anxiety and discomfort, while also facilitating a safe and efficient procedure in the outpatient setting. Ideally, sedative agents have anxiolytic, amnestic, and analgesic properties while maintaining cardiopulmonary stability. The medications used should allow for rapid onset of action, as well as a quick recovery, with minimal side effects.

Several pharmacologic agents are frequently used for conscious sedation in the oral surgery practice. These medications often include midazolam, fentanyl, ketamine and propofol, either alone or in conjunction with one another. While propofol and fentanyl have proved to be efficacious agents for use in intravenous sedation, they are not without associated side effects. Propofol has the potential to cause a quick progression from conscious sedation to general anesthesia, with the undesired effect of associated cardiovascular and respiratory depression. Decreased respiratory drive, hypotension, and dose-dependent bradycardia are often seen with opioid analgesics such as fentanyl.1,2 Ketamine can cause emergence delirium, increased salivation and pulmonary secretions, tachycardia, and post-operative nausea and vomiting (PONV).

Midazolam is a benzodiazepine that is an attractive agent for intravenous sedation due to its sedative, amnestic, and hypnotic properties. In addition, it is associated with very minimal cardiovascular and respiratory changes. However, midazolam lacks significant analgesic effects, and therefore is routinely used in conjunction with additional agents when used for procedural sedation. Though several studies have explored the use of midazolam as a sole anesthetic, very high doses are required for deep sedation. This can lead to dose-dependent respiratory depression, prolonged emergence and longer recovery time.

Dexmedetomidine (Precedex, Hospira, Inc., Lake Forest, IL) is a highly selective alpha2-adrenergic agonist that possesses hypnotic, sedative, anxiolytic, and analgesic properties. It is currently approved for use as a sedative agent in ICU patients, and has been proven a safe and effective agent for use during procedural sedation. In the central nervous system, the primary site of action of dexmedetomidine is the locus ceruleus, resulting in a level of sedation similar to natural sleep, associated with fast and easy arousal. It demonstrates relative hemodynamic stability with little effect on respiratory depression. Unlike propofol and fentanyl, dexmedetomidine's lack of adverse effects on respiration makes it an attractive agent for use during intravenous sedation in the oral and maxillofacial surgery practice.

Several studies involving dexmedetomidine exist in the oral and maxillofacial surgery literature. Dexmedetomidine has been compared as a substitute for midazolam, as well as propofol, in conscious sedation by several authors. For third molar surgery, dexmedetomidine was noted to preserve the respiratory rate and oxygen saturation throughout operation and recovery periods. Fan et al also found no significant differences in respiratory rate when comparing the two agents for conscious sedation. In comparison to midazolam, Ryu et al reported safe sedation without airway compromise and minimal effects on the respiratory system.

Dexmedetomidine also possesses sympatholytic properties, and is commonly associated with a dose-dependent decrease in both heart rate and blood pressure.4,9 Taniyama et al compared dexmedetomidine to propofol for intravenous sedation for minor oral surgical procedures. They found that dexmedetomidine lead to significant hemodynamic changes during the initial loading infusion. An initial increase in blood pressure was seen, followed by a significant decrease in both systolic and diastolic blood pressure, as well as heart rate. These variations are attributed to the fact that dexmedetomidine does not have selectivity for alpha-2A versus alpha-2B receptors. While alpha-2A receptors are found in the CNS and are therefore responsible for the analgesic and sedative effects of the drug, alpha-2B receptors are found in vascular smooth muscle and thereby mediate the hypertensive effects of high doses of dexmedetomidine. Because of this, initial loading doses of dexmedetomidine may be associated with a transient increase in blood pressure, followed by an overall reduction in blood pressure and heart rate from baseline. Hall et al reported that dexmedetomidine demonstrated a decrease in heart rate from baseline between 16 and 18%, and a decrease in blood pressure of 10 to 20%.15 However, in some studies, similar biphasic changes were not observed, possibly due to the use of a lower dosage of dexmedetomidine.

Aside from dose-dependent depression of the cardiovascular system, dexmedetomidine has been associated with minimal to no amnesic effects. One other possible disadvantage of dexmedetomidine as a sedative agent for in-office procedures is the increased postoperative recovery time. Peak sedative effects of the drug occur approximately 90-105 minutes after administration, continuing to as much as 180 minutes. This may necessitate post-operative observation periods of increased duration. Intravenously administered dexmedetomidine has a distribution half-life of 6 minutes and an elimination half-life of 2 hours. It undergoes biotransformation in the liver and is excreted primarily in the urine.

The purpose of this study is to measure the relative efficacy (sedation, analgesia, operating conditions, and patient satisfaction) and safety (hemodynamic and respiratory changes) of dexmedetomidine and midazolam compared to the traditional combination of midazolam, fentanyl, and propofol in office based intravenous sedation for extraction of third molars.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have 3-4 partial or full bony impacted third molars requiring surgical extraction
* ASA Class I or II
* English-speaking and Spanish-speaking subjects

Exclusion Criteria:

* ASA Class III or higher
* Patients taking alpha-2 agonists or benzodiazepines
* Allergy or drug reaction to any of the drugs used in this study (benzodiazepines, opioids, propofol, alpha-2 agonists, NSAIDs, local anesthetic)
* BMI greater than 30
* History of or current substance abuse or alcoholism
* History of mood-altering medications, tranquilizers, or antidepressants.
* Pregnant females

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roback MG, Wathen JE, MacKenzie T, Bajaj L. A randomized, controlled trial of i.v. versus i.m. ketamine for sedation of pediatric patients receiving emergency department orthopedic procedures. Ann Emerg Med. 2006 Nov;48(5):605-12. doi: 10.1016/j.annemergmed.2006.06.001. Epub 2006 Aug 14. PMID 17052563
- [Background] Roback MG, Wathen JE, Bajaj L, Bothner JP. Adverse events associated with procedural sedation and analgesia in a pediatric emergency department: a comparison of common parenteral drugs. Acad Emerg Med. 2005 Jun;12(6):508-13. doi: 10.1197/j.aem.2004.12.009. PMID 15930401
- [Background] Barone CP, Pablo CS, Barone GW. Postanesthetic care in the critical care unit. Crit Care Nurse. 2004 Feb;24(1):38-45. No abstract available. PMID 15007891
- [Background] Eberl S, Preckel B, Bergman JJ, Hollmann MW. Safety and effectiveness using dexmedetomidine versus propofol TCI sedation during oesophagus interventions: a randomized trial. BMC Gastroenterol. 2013 Dec 30;13:176. doi: 10.1186/1471-230X-13-176. PMID 24377675
- [Background] Parworth LP, Frost DE, Zuniga JR, Bennett T. Propofol and fentanyl compared with midazolam and fentanyl during third molar surgery. J Oral Maxillofac Surg. 1998 Apr;56(4):447-53; discussion 453-4. doi: 10.1016/s0278-2391(98)90710-8. PMID 9541344
- [Background] Jun NH, Shim JK, Choi YS, An SH, Kwak YL. Effect of ketamine pretreatment for anaesthesia in patients undergoing percutaneous transluminal balloon angioplasty with continuous remifentanil infusion. Korean J Anesthesiol. 2011 Oct;61(4):308-14. doi: 10.4097/kjae.2011.61.4.308. Epub 2011 Oct 22. PMID 22110884
- [Background] Ustun Y, Gunduz M, Erdogan O, Benlidayi ME. Dexmedetomidine versus midazolam in outpatient third molar surgery. J Oral Maxillofac Surg. 2006 Sep;64(9):1353-8. doi: 10.1016/j.joms.2006.05.020. PMID 16916668
- [Background] Fan TW, Ti LK, Islam I. Comparison of dexmedetomidine and midazolam for conscious sedation in dental surgery monitored by bispectral index. Br J Oral Maxillofac Surg. 2013 Jul;51(5):428-33. doi: 10.1016/j.bjoms.2012.08.013. Epub 2012 Oct 8. PMID 23058230
- [Background] Makary L, Vornik V, Finn R, Lenkovsky F, McClelland AL, Thurmon J, Robertson B. Prolonged recovery associated with dexmedetomidine when used as a sole sedative agent in office-based oral and maxillofacial surgery procedures. J Oral Maxillofac Surg. 2010 Feb;68(2):386-91. doi: 10.1016/j.joms.2009.09.107. PMID 20116712
- [Background] Cheung CW, Ying CL, Chiu WK, Wong GT, Ng KF, Irwin MG. A comparison of dexmedetomidine and midazolam for sedation in third molar surgery. Anaesthesia. 2007 Nov;62(11):1132-8. doi: 10.1111/j.1365-2044.2007.05230.x. PMID 17924894
- [Background] Cheung CW, Ng KF, Liu J, Yuen MY, Ho MH, Irwin MG. Analgesic and sedative effects of intranasal dexmedetomidine in third molar surgery under local anaesthesia. Br J Anaesth. 2011 Sep;107(3):430-7. doi: 10.1093/bja/aer164. Epub 2011 Jun 16. PMID 21685111
- [Background] Bhana N, Goa KL, McClellan KJ. Dexmedetomidine. Drugs. 2000 Feb;59(2):263-8; discussion 269-70. doi: 10.2165/00003495-200059020-00012. PMID 10730549
- [Background] Jaakola ML. Dexmedetomidine premedication before intravenous regional anesthesia in minor outpatient hand surgery. J Clin Anesth. 1994 May-Jun;6(3):204-11. doi: 10.1016/0952-8180(94)90060-4. PMID 7914737
- [Background] Nooh N, Sheta SA, Abdullah WA, Abdelhalim AA. Intranasal atomized dexmedetomidine for sedation during third molar extraction. Int J Oral Maxillofac Surg. 2013 Jul;42(7):857-62. doi: 10.1016/j.ijom.2013.02.003. Epub 2013 Mar 14. PMID 23497981
- [Background] Smiley MK, Prior SR. Dexmedetomidine sedation with and without midazolam for third molar surgery. Anesth Prog. 2014 Spring;61(1):3-10. doi: 10.2344/0003-3006-61.1.3. PMID 24697819
- [Background] Ryu DS, Lee DW, Choi SC, Oh IH. Sedation Protocol Using Dexmedetomidine for Third Molar Extraction. J Oral Maxillofac Surg. 2016 May;74(5):926.e1-7. doi: 10.1016/j.joms.2015.12.021. Epub 2016 Jan 7. PMID 26850877
- [Background] Taniyama K, Oda H, Okawa K, Himeno K, Shikanai K, Shibutani T. Psychosedation with dexmedetomidine hydrochloride during minor oral surgery. Anesth Prog. 2009 Autumn;56(3):75-80. doi: 10.2344/0003-3006-56.3.75. PMID 19769420
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Background] Chanques G, Payen JF, Mercier G, de Lattre S, Viel E, Jung B, Cisse M, Lefrant JY, Jaber S. Assessing pain in non-intubated critically ill patients unable to self report: an adaptation of the Behavioral Pain Scale. Intensive Care Med. 2009 Dec;35(12):2060-7. doi: 10.1007/s00134-009-1590-5. PMID 19697008

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol Group | Dexmedetomidine Group
Started | 69 | 75
Completed | 67 | 74
Not Completed | 2 | 1
Not completed — Under-sedation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol Group | Dexmedetomidine Group | Total
Number analyzed (Participants) | 69 | 75 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (2.7) | 21.4 (2.5) | 21.4 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 46 | 96
  Male | 19 | 29 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Race/Ethnicity Not Collected Population: Race/Ethnicity Not Collected
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (5.2) | 26.1 (5.4) | 25.7 (5.4)
Number of Impactions [Mean (Standard Deviation); unit: Impacted Teeth] | 3.6 (0.5) | 3.6 (0.5) | 3.6 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Events Requiring Intervention
Description: To compare the groups regarding the number of respiratory events requiring intervention, described as: Chin lift/jaw thrust, Tongue thrust, Yankauer suctioning, Positive pressure oxygen administration, Placement of an oral or nasal airway.
Time Frame: During surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
Participants | 17 | 2

2. Secondary Outcome: Reaction to Administration of Local Anesthesia
Description: To compare the groups regarding movement of the patient during the first injection of local anesthesia during the IVS at time of injection measured using the Behavioral Pain Scale - Non-Intubated patients.
  The minimum value is 3 and the maximum value is 12. Higher scores mean a worse outcome (i.e., more pain and movement on injection)
Time Frame: During the first injection of local anesthesia during surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
score on a scale | 3.9 (1.5) | 4.2 (1.4)

3. Secondary Outcome: Patient Satisfaction
Description: Visual Analog Scale was used to measure overall satisfaction with the IV sedation and memory of the procedure.
  The minimum score is 0 (not satisfied at all) to a maximum score of 100 (completely satisfied).
  A higher score is a better outcome.
Time Frame: 30 minutes following surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
score on a scale | 93.5 (10.1) | 86.6 (22.0)

4. Secondary Outcome: Surgeon Satisfaction - Survey
Description: Surgeon satisfaction was measured by the surgeon grading the "Operating Conditions" scale.
  The minimum value was 0 and the maximum was 3. 0=very poor, 1=poor, 2=fair, 3=good
Time Frame: 15 minutes following surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
score on a scale | 2.8 (0.5) | 2.9 (0.4)

5. Secondary Outcome: Cooperation Scale
Description: Surgeon satisfaction is measured by the Cooperation Scale. Minimum score of 0 and maximum of 9. Higher indicates a worse outcome (i.e., discomfort and movement)
Time Frame: 15 minutes following surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
score on a scale | 2.07 (1.95) | 1.47 (1.68)

6. Secondary Outcome: Hemodynamic Stability - Heart Rate
Description: To compare the differences in hemodynamic stability using a D/M combination compared to the MFP combination. (In this study, a deviation from baseline of both the blood pressure and heart rate by 20% or greater will be considered clinically significant)
  a. Change in heart rate (change ≥ 20 BPM)
Time Frame: During the procedure, up to 40 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
beats per minute | 77 (14.20) | 62 (12.28)

7. Secondary Outcome: Hemodynamic Stability - Blood Pressure
Description: To compare the differences in hemodynamic stability using a D/M combination compared to the MFP combination. (In this study, a deviation from baseline by 20% or greater will be considered clinically significant)
  a. Change in blood pressure (NIBP) (change ≥ 20%) Blood pressure is presented as mean arterial pressure
Time Frame: During the procedure, up to 40 minutes
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
mm Hg | 78 (12.4) | 88 (9.25)

8. Secondary Outcome: Respiratory Depression - Respiratory Rate
Description: To assess whether a D/M combination leads to a significant change in respiratory depression compared to the MFP combination.
  a. Change in respiratory rate (change ≥ 20%)
Time Frame: During the procedure, up to 40 minutes
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
breaths per minute | 18 (4.38) | 18 (3.61)

9. Secondary Outcome: Respiratory Depression - Oxygen Saturation
Description: To assess whether a D/M combination leads to a significant change in respiratory depression compared to the MFP combination.
  a. Change in arterial oxygen saturation (as measured by pulse oximeter) i. number of events of ≤92%
Time Frame: During the procedure, up to 40 minutes
Measure: Mean (Standard Deviation); unit: Saturation percent
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
Saturation percent | 98.7 (1.03) | 98.9 (0.37)

10. Secondary Outcome: Postoperative Recovery Time - Duration of Procedure
Description: To assess whether a D/M combination increases postoperative recovery time when compared the MFP combination.
  a. Duration of procedure will be recorded
Time Frame: During the procedure, up to 40 minutes
Measure: Mean (Standard Deviation); unit: MINUTES
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
MINUTES | 24.2 (13.9) | 22.1 (8.8)

11. Secondary Outcome: Postoperative Recovery Time - Ambulation
Description: To assess whether a D/M combination increases postoperative recovery time when compared the MFP combination.
  a. Time to ambulation (to recovery room) will be recorded
Time Frame: After the procedure until ambulation, up to 20 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
minutes | 10.8 (8.6) | 11.6 (6.4)

12. Secondary Outcome: Postoperative Recovery Time - Time to Discharge
Description: To assess whether a D/M combination increases postoperative recovery time when compared the MFP combination.
  a. Time to discharge or "virtual discharge" (comparative statistic) - Aldrete score of ≥ 9 or pre-procedure score is met The minimum score is 0 and the maximum score is 10. A higher score indicates wakefulness, hemodynamically stable, and able to ambulate.
  ii. All subjects are required to stay a minimum of 30 minutes after the end of the procedure. Therefore, at least two postoperative vital sign readings will be obtained. If the subject meets discharge criteria prior to 30 minutes, this time will be the "virtual discharge" time
Time Frame: After the procedure until discharge, up to 45 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Propofol Group | Dexmedetomidine Group
Number analyzed (Participants) | 67 | 74
minutes | 26.5 (14.9) | 29.9 (12.9)

ADVERSE EVENTS:
Time Frame: 90 minutes
Arm/Group | Propofol Group | Dexmedetomidine Group
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/74
Other Adverse Events (participants affected / at risk) | 0/67 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03255824/Prot_SAP_000.pdf